CLINICAL TRIAL: NCT01399398
Title: PET Imaging of CB1 Receptors Using [11C]SD5024
Brief Title: Imaging of CB1 Receptors Using (11C)SD5024
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 110202; 11-M-0202
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2013-12-18

CONDITIONS: Healthy
Keywords: Brain Scan; Kinetic Analysis; Healthy Subjects; Healthy Volunteer; HV
MeSH Terms: interventions — Vascular Access Devices; Blood Specimen Collection

INTERVENTIONS:
Procedure: Brain Scan-PET
Procedure: Brain Scan-MRI
Procedure: Arterial Line
Procedure: Venous Line
Procedure: Blood Sampling

SUMMARY:
Background:

- The cannabinoid type 1 (CB1) receptor is a protein found on some brain cells. It may play a role in obesity or some psychiatric disorders such as schizophrenia. Imaging studies like positron emission tomography (PET) can show where CB1 receptors are located. A new radioactive chemical, 11C-SD5024, may be able to show these receptors more clearly than previous radioactive chemicals. Better images of CB1 receptors in the brain may help improve our understanding of obesity and psychiatric disorders. This information may lead to better treatments.

Objectives:

- To test how well a new radioactive chemical, 11C-SD5024, is taken up by the brain during imaging studies.

Eligibility:

- Healthy volunteers between 18 and 50 years of age who are able to have positron emission tomography scans.

Design:

* All participants will be screened with a physical exam, medical history, and blood tests.
* Participants will be in one of three groups for the study. Each group will receive 11C-SD5024 and have a different set of imaging studies.
* Group 1 will have a magnetic resonance imaging (MRI) scan and PET scan of the brain. They will also have blood and urine tests.
* Group 2 will have a whole-body PET scan, as well as blood and urine tests.
* Group 3 will have an MRI scan of the brain, followed by two PET scans of the brain. They will also have blood and urine tests. The two PET scans can happen on the same day or on two different days.

DETAILED DESCRIPTION:
The cannabinoid type 1 (CB(1)) receptor is one of the most abundant G protein-coupled receptors in the brain (Matsuda et al 1990). It is found on glutamatergic, dopaminergic, and gamma aminobutyric acid (GABA)-ergic synaptic terminals and mediates the effects of endocannabinoids (ECs), which suppresses the release of neurotransmitters. The CB(1) receptor is a target for drug therapy, including the use of a CB(1) receptor antagonist as an appetite suppressant. Our laboratory recently developed a promising positron emission tomography (PET) ligand for the CB(1) receptor: [(11)C]SD5024 (Donohue et al 2008a).

Previous studies from our laboratory used two PET ligands to image CB(1) receptors (11)C-MePPEP and (18)F-FMPEP-d(2) (Yasuno et al 2008; Donohue et al 2008b) and found that the latter provides more accurate and precise measurement. We also found that clearance of (11)C-MePPEP from brain was too slow for (11)C-labeling (Terry et al 2010). Although we are currently using [(18)F]FMPEP-d(2) , the major disadvantage of the current radioligand is that it washes out slowly from the brain, and accurate quantitation requires relatively fast washout. If [(11)C]SD5024 is amenable to quantitation in human subjects, then it may prove to be a useful ligand for studying potential pathophysiological changes of this receptor.

The purpose of this protocol is (1) to perform brain imaging using [(11)C]SD5024 in healthy volunteers to characterize brain uptake and distribution; (2) to perform whole body PET studies in healthy volunteers in order to estimate radiation absorbed doses for [(11)C]SD5024; and (3) to perform brain test-retest studies in healthy volunteers to further examine how precise measurements of receptor binding are, and to determine optimal parameters for future experiments using [(11)C]SD5024.

Successful development of a PET radioligand to image CB1 receptors has the potential to significantly impact our understanding and clinical management of neuropsychiatric (eg, schizophrenia) (Eggan et al 2008) and metabolic (eg, obesity) (Gazzerro et al 2007) disorders. Future experiments would include studies of relevant neuropsychiatric disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy control subjects aged 18 50 whose medical history, physical exam, electrocardiogram (ECG), and laboratory test results are within normal limits within one year of the PET scan will be eligible to participate.

EXCLUSION CRITERIA:

Any recent or past history of psychiatric illness or severe systemic disease based on history and physical exam.

Serious medical illness likely to modify brain anatomy and/or physiology (head trauma, past brain surgery, neurological disorders such as epilepsy, Parkinson disease, and psychiatric disorders such as schizophrenia and depression)

Any current substance or alcohol abuse, with the exception of nicotine.

Positive urine toxicology screen

Radiation exposure from participation in other research protocols in the last year such that the additional radiation exposure from this protocol would exceed annual limits.

Pregnant or breastfeeding.

Claustrophobia (applies to Parts 1 and 3 only).

Metallic (ferromagnetic) implants, including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, shrapnel fragments, and possible small metal fragments in the eye (applies to Parts 1 and 3 only).

Unable to lie flat on back for up to 2.5 hours.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-06-22; Primary Completion 2013-12-18 (Actual); Study Completion 2013-12-18 (Actual)

PRIMARY OUTCOMES:
For the PET scans, we will measure the regional densities of cannabinoid 1 receptors as distribution volume (VT). Distribution volume is the ratio at equilibrium of brain uptake to the concentration of parent radioligand in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Burger C, Buck A. Requirements and implementation of a flexible kinetic modeling tool. J Nucl Med. 1997 Nov;38(11):1818-23. PMID 9374364
- [Background] Cloutier RJ, Smith SA, Watson EE, Snyder WS, Warner GG. Dose to the fetus from radionuclides in the bladder. Health Phys. 1973 Aug;25(2):147-61. doi: 10.1097/00004032-197308000-00009. No abstract available. PMID 4784245
- [Background] Donohue SR, Pike VW, Finnema SJ, Truong P, Andersson J, Gulyas B, Halldin C. Discovery and labeling of high-affinity 3,4-diarylpyrazolines as candidate radioligands for in vivo imaging of cannabinoid subtype-1 (CB1) receptors. J Med Chem. 2008 Sep 25;51(18):5608-16. doi: 10.1021/jm800329z. PMID 18754613